CLINICAL TRIAL: NCT06366100
Title: Dissemination, Acceptability and Adaptation Study of Two Transdiagnostic Psychological Interventions Based on Emotional Regulation (ER) for the Treatment of Alcohol Addiction: Dialectical Behavioral Therapy(DBT) and Unified Protocol (UP)
Brief Title: Implementation of Two Transdiagnostic Interventions Based on Emotional Regulation (DBT and UP) for Alcohol Addiction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Collaborators: Ministerio de Sanidad, Servicios Sociales e Igualdad (Other Government)
Responsible Party: Principal Investigator, María Vicenta Navarro Haro, Associate Professor, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023I060
Record Dates: First submitted 2024-04-02; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Implementation Science
Keywords: Implementation science; Alcohol addiction; Transdiagnostic interventions; Dialectical Behavior Therapy; Unified Protocol
MeSH Terms: conditions — Alcoholism | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two groups in parallel for the duration of the study. The specific design is an reverse counterbalanced (ABBA) intrasubject experimental study where participants will be randomly assigned to first (and then the other) receive DBT-SUD or UP online training in the phase 1 of the study, and randomly assigned to first implement DBT-SUD or UP intervention in the phase two. A balanced randomization (1:1) will be conducted in order to eliminate possible biases and ensure equivalence between groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dialectical Behavior Therapy for Substance Use Disorders (DBT-SUD) (Experimental): In the first phase of the study, a three-day workshop (20 hours) online training on DBT-SUD intervention will be provided to professionals. In the second phase, participants will implement DBT-SUD in group that will consist of applying the skills training mode of DBT for 3 months (12-14 sessions, two hours each). Regarding the specific contents, they will be based on the program published by Maffei´s team (DBT certified trainer and therapist in Italy), which has shown good results in improving the severity and frequency of alcohol use and emotional dysregulation with a 3-month program. Four modules of the skills training program will be applied: mindfulness, distress tolerance, skills to deal with addiction and emotional regulation skills. A self-management and rehabilitation module will be also included.
  Interventions: Behavioral: Dialectical Behavior Therapy for Substance Use Disorder (DBT-SUD)
- Unified Protocol (UP) (Experimental): In the first phase of the study, a a three-day workshop (20 hours) online training on UP intervention will be provided to professionals. In the second phase, participants will implement the UP program that will consist of 8 treatment modules that include training in 5 core skills of emotional regulation: mindfulness training, cognitive flexibility, identification/oppositional behavior of emotional behaviors, interoceptive exposure and emotional exposure. Our team has adapted the UP to be implemented in 12 group sessions, one per week, lasting 2 hours, in specialized mental health care services of the national health system. Additional recommendations to adapt UP to alcohol addiction will be included.
  Interventions: Behavioral: Unified Protocol (UP)

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy for Substance Use Disorder (DBT-SUD) — In phase 1, DBT online training will consist of the following contents:
  Block 1
  1.1. Introduction to the key concepts 1.2. DBT-SUD program 1.3. Why DBT for alcohol addiction? 1.4. Proposed content for the group intervention.
  Block 2
  2.1. DBT skills training modules
  In phase 2, DBT-SUD intervention will consist of about the following sessions:
  GOALS OF SKILLS TRAINING AND MINDFULNESS:
  S1: Goals of skills training; Observing, Describing and Participating
  S2: Non-judgmentally, One-mindfulness, Effectively
  DISTRESS TOLERANCE:
  S3: Crisis Survival skills
  S4: Crisis Survival and Radical Acceptance
  ADDICTION SKILLS:
  S5: Dialectical Abstinence.
  S6: Clear Mind
  S7: Burning Bridges-Building New Bridges
  S8: Community Reinforcement
  EMOTIONAL REGULATION:
  S9: Identifying emotions and model of emotion
  S10: Check the facts. Opposing Action
  S11: Problem Solving. Reducing vulnerability
  S12: Self-management and rehabilitation
  Arms: Dialectical Behavior Therapy for Substance Use Disorders (DBT-SUD)
Behavioral: Unified Protocol (UP) — In phase 1, the UP training will have following contents:
  Block 1
  1.1. Introduction to key concepts 1.2. Why UP for alcohol addiction? 1.3. Dimensional assessment and case formulation. 1.4. Main characteristics of UP
  Block 2
  2.1. Modules of UP
  In phase 2, UP intervention will consist of:
  MOTIVATION:
  S1: Motivation enhancement for treatment
  UNDERSTANDING EMOTIONS:
  S2: Understanding and model of emotions S3: Tracking emotional responses
  MINDFULNESS:
  S4: Emotion awareness
  COGNITIVE FLEXIBILITY:
  S5: Cognitive reappraisal to increase thinking flexibility
  EMOTION DRIVEN BEHAVIORS:
  S6: Emotional avoidance S7: Emotion-driven behaviors and alternative action
  AWARENESS AND TOLERANCE:
  S8: Tolerance of physical sensations
  EMOTIONAL EXPOSURE:
  S9: Interoceptive and situational emotion exposure S10: Exposure practice
  RELAPSE PREVENTION:
  S11: Relapse prevention S12: Review of progress
  Arms: Unified Protocol (UP)

SUMMARY:
The aim of this study is to evaluate the dissemination and implementation process of two transdiagnostic psychological interventions (Dialectical Behavioral Therapy for Substance Use Disorders-DBT-SUD and Unified Protocol-UP) to treat alcohol addiction by mental health practitioners in the Spanish National Health System. The main questions this study aims to answer are:

Are there differences before and after receiving DBT-SUD and UP training in the attitudes toward evidence-based psychological treatments (EBPTs), level of burnout and organizational climate and readiness to implement the interventions in mental health practitioners working with alcohol addiction?

What is the degree of acceptability and intention to use the interventions in clinical practice with people with alcohol addiction of the practitioners after each training (DBT-SUD and UP)?

In what degree the implementation outcomes (adoption, reach, appropriateness, feasibility, fidelity, sustainability) will be achieved by the practitioners implementing DBT-SUD and UP in clinical practice?

What are the main barriers and facilitators that practitioners will encounter during the process of implementing DBT-SUD and UP in clinical practice?

What variables will predict a successful implementation considering previous characteristics of the professionals and the organizational outcomes?

The study comprises two phases. In the first phase, mental health professionals working on addiction services of the Spanish National Health System will be randomly assigned to receive training in one intervention and then the other (DBT-SUD and UP) and will be evaluated before and after each training. In the second phase, participants will be randomly assigned to implement one intervention first and then the other in their workplaces with people with alcohol addiction and will be also assessed before and after the implementation. Qualitative and quantitate outcome measures will be analyzed using a Mixed- Methods-Design.

DETAILED DESCRIPTION:
Alcohol addiction is among the most frequent mental health problems in Spain, affecting more than 4% of the general population and it accounts for around 35% of admissions to outpatient services of Spanish National Health System (NHS). Alcohol addiction has significant morbidity and mortality, and several comorbidities that limit the effectiveness of psychological treatments. The scientific literature suggests that emotional dysregulation is one of the most important determinants of craving and relapse, therefore may represent a promising target for improving psychological treatments for alcohol addiction. Recently, different transdiagnostic psychological treatments have been focused on the etiological and maintenance mechanisms underlying different disorders, providing a comprehensive model to treat emotion dysregulation. From this perspective, alcohol use has been considered a maladaptive behavior to regulate aversive emotional states. DBT and UP are two examples of transdiagnostic treatments with good efficacy and effectiveness results to treat emotion dysregulation and have shown preliminary effectiveness to treat alcohol addiction. Research studies on psychological treatments have traditionally focused on the efficacy of evidence-based interventions. However, there is a major problem in translating these treatments into the clinical practice. Because research on dissemination and implementation is a relatively new area of study in the addictions field, little is known about how to optimize the implementation of evidence-based psychological treatment. One of the main barriers encountered in the implementation of psychological interventions for alcohol addiction is the inadequate training of professionals. With regard to facilitators, providers' familiarity with the interventions, perception of their effectiveness, and attitudes toward them have been found to be associated with the likelihood of success in treatment implementation.

In this study, two sequential phases are proposed. The first phase aims to evaluate the effect of the dissemination of two treatments (DBT-SUD and UP) on the attitudes, readiness to change, acceptability and intention to use these interventions in mental health professionals, as well as to explore information on the adaptation of both interventions to real contexts of public addiction settings. The participants in phase 1 will be at least 160 mental health professionals (psychiatrist, psychologist and nurse) who work in the Spanish NHS drug addiction services of Aragón, Valencia and Catalonia regions and are treating people with alcohol addiction. In this phase 1, after they provide informed consent, participants will be randomized assigned to receive online training in one intervention and then the other (DBT-SUD and UP; the content of these trainings can be consulted in the intervention section) and will complete a series of questionnaires before and after each training. In addition to the battery of questionnaires (they are described in the outcome measures section), to collect qualitative information, participants will be given the possibility to participate in small focus groups. The questions included in the focus group interviews will explore the acceptability and intention to use both interventions (DBT and UP) as well as possible adaptations that would be needed to implement them in clinical practice.

The second phase aims to evaluate variables regarding implementation (i.e. barriers, adoption, adequation, fidelity) of the interventions. The main purpose of this phase is to promote an adequate implementation of transdiagnostic interventions in the reality of addiction services of the NHS. In this phase 2 of the study, it was expected to recruit at least 20% of the professionals trained in phase 1. Participants will be randomly assigned to implement one of the interventions first, and then the other (DBT-SUD or UP). Quantitative measures will be administered before, during and after the implementation process. Professionals may voluntarily participate in small discussion groups. The following variables are proposed to be evaluated during this phase: 1) acceptability; 2) adoption and reach; 3) appropriateness; 4) feasibility; 5) fidelity; 6) barriers and facilitators of implementation. The implementation of DBT-SUD and UP interventions will be done in a group format and will last around 3 months in a weekly basis (between 12-14 sessions, two hours per session). The interventions will be adapted according to the context in which they are applied following the feedback collected by the professionals. The DBT-SUD program will consist of applying the DBT skills training. The specific contents will be based on Maffei´s team adaptations of DBT for alcohol addiction, which include emotion regulation skills, distress tolerance, mindfulness (present moment awareness) and addiction skills and has shown good results in improving the severity and frequency of alcohol consumption and emotional dysregulation with a 3-month program. The UP will consist of 8 treatment modules that include training in 5 core emotional regulation skills: mindfulness training, cognitive flexibility, identification/oppositional behavior of emotional behaviors, interoceptive exposure, and emotional exposure. The content of the intervention will be based on previous recommendations for the adequate implementation of the UP in substance use disorders. To guarantee implementation of the interventions, supervisions by the experts will be carried out session by session with the aim of evaluating treatment fidelity and help practitioners overcome barriers during the implementation process.

ELIGIBILITY:
Phase 1:

Inclusion Criteria:

* Be at least 18 years of age
* Mental health professional (psychologist, psychiatrist, nurse) currently working in an addiction treatment service
* Agree to receive training in DBT and UP programs
* Understand Spanish
* Accept informed consent

Exclusion Criteria:

* Not being interested in receiving training in emotional regulation interventions
* Not including in their functions, the psychological treatment of people with alcohol addiction
* Not having an Internet connection to be able to connect to the training sessions

Phase 2:

Inclusion criteria:

* Be at least 18 years of age
* Psychologists currently working in an addiction treatment service
* Have received training in DBT and UP interventions in phase 1
* Accept the implementation of any of the 2 interventions and the supervision during the implementation
* Understand the Spanish language
* Accept the informed consent

Exclusion criteria:

* Not being interested in implementing and/or receiving supervision in the interventions
* Not including in their functions, the psychological treatment of people with alcohol addiction
* Not having an Internet connection to be able to connect to the supervision sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability and Intention to Use Survey | Phase 1: Last session of DBT and UP trainings; up to 3 weeks for each training (3 weekly sessions of 6-7 hours each); Phase 2: Last session of DBT or UP implementation (3 months, 12-14 weeks for each intervention)
  This 9-item instrument is based on the Theoretical Framework of Acceptability (TFA) and assesses acceptability and unifies approaches into a single theoretical framework. The model is composed of seven constructs: Affective attitude; Burden; Ethics; Consistency of intervention; Opportunity costs; Perceived efficacy and Self-efficacy. This questionnaire was created ad hoc in Spanish language by the authors of the instrument and adds two more items reflecting general acceptability and intention to use the intervention in the future.
Measures of Acceptability, Appropriateness and Feasibility of the intervention (AIM, IAM & FIM) | Phase 1: After DBT and UP trainings; last session of training: up to 3 weeks for each training (3 weekly sessions of 6-7 hours each); Phase 2: Last session of DBT or UP implementation (3 months, 12-14 weeks for each intervention)
  This is a 12-item instrument with three scales (acceptability, appropriateness and feasibility) and contains statements about the intervention to be measured. These measures could be used independently or together. They will be used together in this study. The instrument presents solid psychometric properties: Cronbach alphas were between .87 and .89 and by subscales alpha were .85 for acceptability, .91 for appropriateness and .89 for feasibility (minimum=0.70 and maximum=0.90 acceptable Cronbach´s alpha scores). The original scale has been back-translated for their correct adaptation to Spanish language.
Normalization MeAsure Development Questionnaire (NoMAD) | Phase 2: Before and after implementation: first and last session of DBT or UP (3 months, 12-14 weeks for each intervention)
  This 12-item questionnaire measures implementation processes from the perspective of professionals directly involved in the implementation of complex interventions in health care. It has four dimensions: coherence of the intervention with daily routine, cognitive participation, collective action of individuals and groups to apply the innovation in daily practice, and reflective monitoring. This instrument was validated for the implementation of complex interventions in primary care, showing adequate psychometric properties. Most values for Cronbach alphas for all four of sub-scales (pooled across site) by time point reached satisfactory thresholds: α ≥ 0.70. The Spanish version will be used, which was developed by the ImpleMentAll partners (https://www.implementall.eu/9-outcomes-and-resources.html#NoMADtranslations).

SECONDARY OUTCOMES:
Copenhagen Burnout Inventory (CBI) | Phase 1: Before & after DBT and UP trainings (first and last session of training; up to 3 weeks for each training); Phase 2: Before and after implementation: first and last session of DBT or UP implementation (3 months, 12-14 weeks for each intervention)
  The 18-item questionnaire is in the public domain for the measurement of burnout syndrome, and is structured in three subdimensions: personal, work-related, and work-related with clients. It presents good internal consistency of the three scales: Cronbach's alpha for total instrument was >.70 and of .90 in the personal dimension, .83 in the work-related dimension and .82 in the dimension related to dealing with clients).
Brief Scale of Understanding Substance Abuse (SUSS) | Phase 1: After DBT and UP trainings (first and last session of training; up to 3 weeks for each training); Phase 2: Before and after implementation: first and last session of DBT or UP implementation (3 months, 12-14 weeks for each intervention)
  This 19-items instrument has statements about the nature and etiology of alcohol and substance abuse disorders and consists of three subscales: disease model, psychosocial model, and eclectic orientation. This scale presents good internal consistency scores for its first two scales: Cronbach's alphas of .86 and .72, respectively, and low score .61 for eclectic orientation subscale (minimum=0.70 and maximum=0.90 acceptable Cronbach´s alpha scores) . The scale has been back-translated for their correct adaptation to Spanish language.
Implementation Climate Scale (ICS) | Phase 1: Before and after DBT and UP trainings (first and last session of training; up to 3 weeks for each training); Phase 2: After implementation: last session of DBT or UP (3 months, 12-14 weeks for each intervention)
  This 18-item measure assesses the degree to which there is a strategic organizational climate that supports the implementation of evidence-based practices. the implementation of evidence-based practices. The implementation climate is defined as the perception of the policies, practices, procedures, and behaviors that are rewarded, supported, and expected to facilitate the effective implementation of EBP. This scale was validated with organizations that implemented substance use disorder treatments and showed good psychometric properties. Cronbach's alpha reliabilities for the subscales and ICS total score ranged from .78-.90, demonstrating strong internal consistency reliability (minimum=0.70 and maximum=0.90 acceptable Cronbach´s alpha scores). To adapt this instrument to Spanish, a back-translation was conducted.
Organizational Readiness for Implementing Change (ORIC) | Phase 1: After DBT and UP trainings (first and last session of training; up to 3 weeks for each training); Phase 2: Before and after implementation: first and last session of DBT or UP (3 months, 12-14 weeks for each intervention)
  This 12-item scale is divided into two main subscales: Commitment to change (i.e., do the intended members of the organization want change?) and Effectiveness of change (i.e., can the members of the organization change?). Cronbach's alpha values were, respectively, 0.91 and 0.89 for the Change Commitment Scale and the Change Efficacy Scale. Spanish version was developed by ImpleMentAll partners (https://www.implementall.eu/9-outcomes-and-resources.html#ORICtranslations).
Evidence-Based Practice Attitudes Scale (EBPAS) | Phase 1: Before and after DBT and UP trainings (first and last session of training; up to 3 weeks for each training); Phase 2: After implementation: last session of DBT or UP (3 months, 12-14 weeks for each intervention)
  This 15-item scale assesses participants' attitudes toward adopting evidence-based practice in four domains: Likelihood of adopting EBP given the requirements to do so, Intuitive appeal of EBP, Openness to new practices, and Perceived divergence of usual practice from EBP. The tool presents an overall scale alpha range of .77-.79 and α range of .78-0.93 for subscales, excluding perceived divergence with somewhat lower reliability: α range of .59-.66 (minimum=0.70 and maximum=0.90 acceptable Cronbach´s alpha scores). This subscale was excluded for this study.
Program sustainability assessment tool (PASAT) | Phase 2: After implementation: last session of DBT or UP (3 months, 12-14 weeks for each intervention)
  This is a 40-item scale of intervention sustainability as reported by the organization's provider and stakeholders. The subscales are: political support, funding stability, stakeholder partnerships, organizational capacity, program evaluation, program adaptation, stakeholder communication, and strategic planning. The average internal consistency of the 8 subscales was .88 and ranged from .79-.92 (minimum=0.70 and maximum=0.90 acceptable Cronbach´s alpha scores) . The Spanish version, developed by the Washington University, St. Louis (US) is available on its official website at: https://sustaintool.org/psat/assess/
Barriers to Implementation Inventory (BTI) | Phase 1: Last session of DBT and UP trainings; up to 3 weeks for each training (3 weekly sessions of 6-7 hours each); Phase 2: Last sesion of DBT or UP implementation (3 months, 12-14 weeks for each intervention)
  The 39-item inventory consists of a list of barriers that teams may encounter when implementing DBT. The obstacles are structured by the following domains: team problems, administrative problems, theoretical/philosophical problems, and structural problems. The validation study of the original scale showed adequate psychometric properties, the internal reliability of the scores was good: Cronbach´s alpha .89 (minimum=0.70 and maximum=0.90 acceptable Cronbach´s alpha scores). However, in this some adjustments of the scale were conducted using the barriers reported by the scientific literature when implementing evidence-based treatments for addiction. The scale has been back-translated for their correct adaptation to Spanish.

CONTACTS AND LOCATIONS:
Overall Officials: María Vicenta Navarro Haro, PhD, Principal Investigator — Universidad de Zaragoza
Locations (1):
- University of Zaragoza, Teruel, Aragon, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carlucci L, Saggino A, Balsamo M. On the efficacy of the unified protocol for transdiagnostic treatment of emotional disorders: A systematic review and meta-analysis. Clin Psychol Rev. 2021 Jul;87:101999. doi: 10.1016/j.cpr.2021.101999. Epub 2021 Mar 9. PMID 34098412
- [Background] Luke DA, Calhoun A, Robichaux CB, Elliott MB, Moreland-Russell S. The Program Sustainability Assessment Tool: a new instrument for public health programs. Prev Chronic Dis. 2014 Jan 23;11:130184. doi: 10.5888/pcd11.130184. PMID 24456645
- [Background] Molinero Ruiz E, Basart Gomez-Quintero H, Moncada Lluis S. Validation of the Copenhagen Burnout Inventory to assess professional burnout in Spain. Rev Esp Salud Publica. 2013 Mar-Apr;87(2):165-79. doi: 10.4321/S1135-57272013000200006. English, Spanish. PMID 23775105
- [Background] Ehrhart MG, Torres EM, Hwang J, Sklar M, Aarons GA. Validation of the Implementation Climate Scale (ICS) in substance use disorder treatment organizations. Subst Abuse Treat Prev Policy. 2019 Aug 23;14(1):35. doi: 10.1186/s13011-019-0222-5. PMID 31443666
- [Background] Ehrhart MG, Aarons GA, Farahnak LR. Assessing the organizational context for EBP implementation: the development and validity testing of the Implementation Climate Scale (ICS). Implement Sci. 2014 Oct 23;9:157. doi: 10.1186/s13012-014-0157-1. PMID 25338781
- [Background] Shea CM, Jacobs SR, Esserman DA, Bruce K, Weiner BJ. Organizational readiness for implementing change: a psychometric assessment of a new measure. Implement Sci. 2014 Jan 10;9:7. doi: 10.1186/1748-5908-9-7. PMID 24410955
- [Background] Aarons GA. Mental health provider attitudes toward adoption of evidence-based practice: the Evidence-Based Practice Attitude Scale (EBPAS). Ment Health Serv Res. 2004 Jun;6(2):61-74. doi: 10.1023/b:mhsr.0000024351.12294.65. PMID 15224451
- [Background] Obert JL, Brown AH, Zweben J, Christian D, Delmhorst J, Minsky S, Morrisey P, Vandersloot D, Weiner A. When treatment meets research: clinical perspectives from the CSAT Methamphetamine Treatment Project. J Subst Abuse Treat. 2005 Apr;28(3):231-7. doi: 10.1016/j.jsat.2004.12.008. PMID 15857723
- [Background] Morris ZS, Wooding S, Grant J. The answer is 17 years, what is the question: understanding time lags in translational research. J R Soc Med. 2011 Dec;104(12):510-20. doi: 10.1258/jrsm.2011.110180. PMID 22179294
- [Background] Ciraulo DA, Barlow DH, Gulliver SB, Farchione T, Morissette SB, Kamholz BW, Eisenmenger K, Brown B, Devine E, Brown TA, Knapp CM. The effects of venlafaxine and cognitive behavioral therapy alone and combined in the treatment of co-morbid alcohol use-anxiety disorders. Behav Res Ther. 2013 Nov;51(11):729-35. doi: 10.1016/j.brat.2013.08.003. Epub 2013 Aug 30. PMID 24055681
- [Background] Peris-Baquero O, Osma J, Gil-LaCruz M, Martinez-Garcia L. Acceptability of and intention to use the Unified Protocol delivered in group format in the Spanish Public Health System. J Eval Clin Pract. 2021 Dec;27(6):1299-1309. doi: 10.1111/jep.13546. Epub 2021 Feb 9. PMID 33565231
- [Background] Maffei C, Cavicchioli M, Movalli M, Cavallaro R, Fossati A. Dialectical Behavior Therapy Skills Training in Alcohol Dependence Treatment: Findings Based on an Open Trial. Subst Use Misuse. 2018 Dec 6;53(14):2368-2385. doi: 10.1080/10826084.2018.1480035. Epub 2018 Jun 29. PMID 29958050
- [Background] Cavicchioli M, Movalli M, Vassena G, Ramella P, Prudenziati F, Maffei C. The therapeutic role of emotion regulation and coping strategies during a stand-alone DBT Skills training program for alcohol use disorder and concurrent substance use disorders. Addict Behav. 2019 Nov;98:106035. doi: 10.1016/j.addbeh.2019.106035. Epub 2019 Jun 25. PMID 31302312
- [Background] Spanish Observatory on Drugs and Addictions. Report 2023. Alcohol, tobacco and illegal drugs in Spain. Madrid: Ministry of Health. Government Delegation for the National Plan on Drugs; 2023. 270 p.
- [Background] Connor JP, Haber PS, Hall WD. Alcohol use disorders. Lancet. 2016 Mar 5;387(10022):988-998. doi: 10.1016/S0140-6736(15)00122-1. Epub 2015 Sep 3. PMID 26343838
- [Background] Schuckit MA. Alcohol-use disorders. Lancet. 2009 Feb 7;373(9662):492-501. doi: 10.1016/S0140-6736(09)60009-X. Epub 2009 Jan 23. PMID 19168210
- [Background] Bullis JR, Boettcher H, Sauer-Zavala S, Barlow DH. What is an emotional disorder ? A transdiagnostic mechanistic definition with implications for assessment , treatment , and prevention. Clin Psychol Sci Pract. 2019;1-19.
- [Background] Gamble SA, Conner KR, Talbot NL, Yu Q, Tu XM, Connors GJ. Effects of pretreatment and posttreatment depressive symptoms on alcohol consumption following treatment in Project MATCH. J Stud Alcohol Drugs. 2010 Jan;71(1):71-7. doi: 10.15288/jsad.2010.71.71. PMID 20105416
- [Background] Sinha R. How does stress lead to risk of alcohol relapse? Alcohol Res. 2012;34(4):432-40. PMID 23584109
- [Background] Ritschel LA, Lim NE, Stewart LM. Transdiagnostic Applications of DBT for Adolescents and Adults. Am J Psychother. 2015;69(2):111-28. doi: 10.1176/appi.psychotherapy.2015.69.2.111. PMID 26160618
- [Background] Anker JJ, Kushner MG, Thuras P, Menk J, Unruh AS. Drinking to cope with negative emotions moderates alcohol use disorder treatment response in patients with co-occurring anxiety disorder. Drug Alcohol Depend. 2016 Feb 1;159:93-100. doi: 10.1016/j.drugalcdep.2015.11.031. Epub 2015 Dec 11. PMID 26718394
- [Background] Cassiello-Robbins C, Southward MW, Tirpak JW, Sauer-Zavala S. A systematic review of Unified Protocol applications with adult populations: Facilitating widespread dissemination via adaptability. Clin Psychol Rev. 2020 Jun;78:101852. doi: 10.1016/j.cpr.2020.101852. Epub 2020 Apr 20. PMID 32360953
- [Background] Valentine SE, Smith AM, Stewart K. A review of the empirical evidence for DBT skills training as a stand-alone intervention. Handb Dialect Behav Ther. 2020;325-58.
- [Background] Gold PB, Glynn SM, Mueser KT. Challenges to implementing and sustaining comprehensive mental health service programs. Eval Health Prof. 2006 Jun;29(2):195-218. doi: 10.1177/0163278706287345. PMID 16645184
- [Background] Herbeck DM, Hser YI, Teruya C. Empirically supported substance abuse treatment approaches: a survey of treatment providers' perspectives and practices. Addict Behav. 2008 May;33(5):699-712. doi: 10.1016/j.addbeh.2007.12.003. Epub 2007 Dec 23. PMID 18207334
- [Background] Thomas CP, Wallack SS, Lee S, McCarty D, Swift R. Research to practice: adoption of naltrexone in alcoholism treatment. J Subst Abuse Treat. 2003 Jan;24(1):1-11. PMID 12646325
- [Background] Barlow DH, Farchione TJ, Fairholme CP, Ellard KK, Boisseau CL, Allen LB, et al. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders. New York: Oxford University Press; 2011.
- [Background] Barlow DH, Farchione TJ, Sauer-Zavala S, Latin HM, Ellard KK, Bullis JR, et al. Unified protocol for transdiagnostic treatment of emotional disorders: Therapist guide. New York, NY: Oxford University Press; 2018.
- [Background] Landa González N, Osma J, Peris-Baquero O. Emotional disorders and comorbidity with addictions. In: Applications of the Unified Protocol for the transdiagnostic treatment of emotional dysregulation. Madrid: Alianza Editorial; 2019.
- [Background] Humphreys, K., Greenbaum, MA., Noke, JM., & Finney, JW. Reliability, validity, and normative data for a short version of the Understanding of Alcoholism Scale. Psychology of Addictive Behaviors, 1996 10(1), 38-44. https://doi.org/10.1037/0893-164X.10.1.38
- [Background] Tage S. Kristensen , Marianne Borritz , Ebbe Villadsen & Karl B. Christensen. The Copenhagen Burnout Inventory: A new tool for the assessment of burnout, Work & Stress, 2005 19:3, 192-207, DOI: 10.1080/02678370500297720
- [Background] De Paul J, Indias S, Arruabarrena I. Adaptation of the Evidence-Based Practices Attitude Scale in Spanish child welfare professionals. Psicothema. 2015;27(4):341-6. doi: 10.7334/psicothema2015.67. PMID 26493571
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Finch TL, Girling M, May CR, Mair FS, Murray E, Treweek S, McColl E, Steen IN, Cook C, Vernazza CR, Mackintosh N, Sharma S, Barbery G, Steele J, Rapley T. Improving the normalization of complex interventions: part 2 - validation of the NoMAD instrument for assessing implementation work based on normalization process theory (NPT). BMC Med Res Methodol. 2018 Nov 15;18(1):135. doi: 10.1186/s12874-018-0591-x. PMID 30442094
- [Background] Lamarche L, Clark RE, Parascandalo F, Mangin D. The implementation and validation of the NoMAD during a complex primary care intervention. BMC Med Res Methodol. 2022 Jun 19;22(1):175. doi: 10.1186/s12874-022-01655-0. PMID 35718763
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Farchione TJ, Fitzgerald HE, Curreri A, Janes AC, Gallagher MW, Sbi S, Eustis EH, Barlow DH. Efficacy of the Unified Protocol for the treatment of comorbid alcohol use and anxiety disorders: Study protocol and methods. Contemp Clin Trials. 2021 Sep;108:106512. doi: 10.1016/j.cct.2021.106512. Epub 2021 Jul 17. PMID 34284152
- [Derived] Navarro-Haro MV, Abanades-Morillo A, Peris-Baquero O, Martinez-Borba V, Crespo-Delgado E, Baquero-Escribano A, Masferrer-Boix L, Osma J. Implementation of two transdiagnostic interventions based on emotional regulation for professionals who treat alcohol addiction in the Spanish mental health system: A multicenter mixed methods pilot study protocol. PLoS One. 2025 May 9;20(5):e0318512. doi: 10.1371/journal.pone.0318512. eCollection 2025. PMID 40344573

DOCUMENTS (1):
  • Informed Consent Form (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/00/NCT06366100/ICF_000.pdf